CLINICAL TRIAL: NCT00298597
Title: Influence of G-CSF and EPO on Associative Learning and Motor Skills
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCSFEPO_01; EudraCT Number 2005-001113-18
Record Dates: First submitted 2006-03-01; First posted 2006-03-02 (Estimated); Last update posted 2009-04-23 (Estimated); Status verified 2007-04

CONDITIONS: Chronic Stroke; Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Granulocyte Colony-Stimulating Factor; Erythropoietin

INTERVENTIONS:
Drug: granulocyte - colony stimulating factor (G-CSF)
Drug: erythropoetin (EPO)

SUMMARY:
In the study we want to prove whether the subcutaneous application of granulocyte-stimulating factor (G-CSF) and erythropoetin (EPO) influence associative learning and/or motor skills of patients, who suffer from chronic stroke or amyotrophic lateral sclerosis. The study hypothesis is that G-CSF and EPO improve associative learning and/or motor skills.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic stroke or amyotrophic lateral sclerosis

Exclusion Criteria:

* leucocytes > 10000/µl
* hematocrit > 48%
* thrombocytes < 150000/µl
* severe rheumatoid arthritis
* severe infection
* severe liver or renal failure
* severe arterial hypertension
* recurrent thromboembolic events
* severe coronary heart disease
* myocardial infarction
* malignant tumor
* leukemia
* peripheral arterial occlusion disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2006-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Learning success in a word learning model
Response time in motor function tests

SECONDARY OUTCOMES:
Response time in a word learning model
Total time and number of keystrokes in motor function tests

CONTACTS AND LOCATIONS:
Overall Officials: Wolf Rüdiger Schäbitz, MD, Principal Investigator — Department of Neurology, University Hospital of Muenster, Germany
Locations (1):
- Department of neurology, University Hospital of Muenster, Münster, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Knecht S, Breitenstein C, Bushuven S, Wailke S, Kamping S, Floel A, Zwitserlood P, Ringelstein EB. Levodopa: faster and better word learning in normal humans. Ann Neurol. 2004 Jul;56(1):20-6. doi: 10.1002/ana.20125. PMID 15236398
- [Background] Schneider A, Kuhn HG, Schabitz WR. A role for G-CSF (granulocyte-colony stimulating factor) in the central nervous system. Cell Cycle. 2005 Dec;4(12):1753-7. doi: 10.4161/cc.4.12.2213. Epub 2005 Dec 27. PMID 16258290
- [Background] Schneider A, Kruger C, Steigleder T, Weber D, Pitzer C, Laage R, Aronowski J, Maurer MH, Gassler N, Mier W, Hasselblatt M, Kollmar R, Schwab S, Sommer C, Bach A, Kuhn HG, Schabitz WR. The hematopoietic factor G-CSF is a neuronal ligand that counteracts programmed cell death and drives neurogenesis. J Clin Invest. 2005 Aug;115(8):2083-98. doi: 10.1172/JCI23559. Epub 2005 Jul 7. PMID 16007267
- [Derived] Floel A, Warnecke T, Duning T, Lating Y, Uhlenbrock J, Schneider A, Vogt G, Laage R, Koch W, Knecht S, Schabitz WR. Granulocyte-colony stimulating factor (G-CSF) in stroke patients with concomitant vascular disease--a randomized controlled trial. PLoS One. 2011;6(5):e19767. doi: 10.1371/journal.pone.0019767. Epub 2011 May 23. PMID 21625426
- [Derived] Duning T, Schiffbauer H, Warnecke T, Mohammadi S, Floel A, Kolpatzik K, Kugel H, Schneider A, Knecht S, Deppe M, Schabitz WR. G-CSF prevents the progression of structural disintegration of white matter tracts in amyotrophic lateral sclerosis: a pilot trial. PLoS One. 2011 Mar 14;6(3):e17770. doi: 10.1371/journal.pone.0017770. PMID 21423758